CLINICAL TRIAL: NCT03746340
Title: The Effects of Different General Anesthetics on Serum Folic Acid and Homocysteine Concentrations in Children
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Other Study IDs: SH9H-2018-T53-2
Record Dates: First submitted 2018-11-08; First posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Anesthetic Toxicity
Keywords: sevoflurane; propofol; Folic Acid
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anesthetic: Sevoflurane Group Propofol Group
  Interventions: Drug: Propofol; Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — Propofol group: intravenous Propofol (2.0mg / kg) for general anesthesia induction, maintained for 30~60s. Continuous intravenous infusion of Propofol (7~8 mg·kg-1·h-1) with a syringe pump maintains a smooth general anesthetic sedative effect.
Drug: Sevoflurane — Sevoflurane group: Inhalation of 1-8% sevoflurane for induction.Then Inhalation of sevoflurane (2.0~2.5Vol%) was maintained

SUMMARY:
The concentration of folic acid and homocysteine in the blood can be used as independent risk factors for a variety of diseases. A sustained decrease in blood folate concentration and an increase in homocysteine concentration can damage vascular endothelial cells, causing varying degrees of neurodevelopmental abnormalities. Many clinical studies have found that anesthetics can affect blood folate and homocysteine concentration, but the effects of sevoflurane and propofol on blood folate and homocysteine concentrations are not clear. Therefore, this study aims to investigate the effects of sevoflurane and propofol on blood folate and homocysteine levels in children.

DETAILED DESCRIPTION:
Retrospective study: Study the medical history of infants and young children (less than 3 years old) who underwent sevoflurane or propofol general anesthesia for more than 3 hours from January 2018 to December 2018, and compare the preoperative and postoperative serum folate changes for retrospective analysis.

Prospective study：Ten infants and young children (less than 3 years old) who underwent general anesthesia from November 7, 2018 to December 31, 2018 in Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine. Inhalation of 1-8% concentration of sevoflurane for general anesthesia induced intubation, followed by sevoflurane 2.0 ~ 2.5 Vol% inhalation maintenance, according to the intraoperative situation to add opioids. Patients maintained a bispectral index (BIS) monitoring between 50 and 60. After induction of general anesthesia in all patients, Serum folate levels were measured before the start of surgery, every 1 hour during surgery, and at the end of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Children under 3 years old who underwent general anesthesia
2. Those who did not participate in other clinical trials within 3 months
3. No acute infectious diseases, systemic diseases
4. The family member of the child agrees to the test and signs the informed consent form.

Exclusion Criteria:

1. Refusal to join the group
2. severe liver and kidney damage
3. Hemodynamic instability (shock, blood pressure drop > 30% of basal blood pressure)
4. Children with egg and milk allergy
5. Children with a family history of malignant hyperthermia

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under 3 years old who underwent general anesthesia
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
levels of folate in the perioperative serum | Change of serum folate levels from the beginning of anesthesia to the end.Serum folate levels were measured at admission, after 1 hours,after 2 hours,after 3 hours.
  a Chemiluminescent Microparticle Folate Binding Protein assay with the ARCHITECT Folate Reagent Kit (Abbott Laboratories, IL, USA) was used to determine serum folate concentrations. Serum folate concentrations were quantified using the ARCHITECT i2000 SR System (Abbott Laboratories).
levels of homocysteine in the perioperative serum | Change of serum homocysteine levels from the beginning of anesthesia to the end.Serum homocysteine levels were measured at admission, after 1 hours,after 2 hours,after 3 hours.
  Serum Hcy concentrations were analyzed by fluorescence polarization immunoassay using the IMx Homocysteine Reagent Pack and IMx Analyzer (Abbott Laboratories).

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jiang, MD,PhD, Principal Investigator — Shanghai Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Ninth People's Hospital , Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China